CLINICAL TRIAL: NCT05732688
Title: Drug-screening in AML at Relapse for Targeted Treatment
Acronym: DARTT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DARTT-1
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: AML
Keywords: AML; Relapse; Drug-screening; Pharmacoscopy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacoscopy (Experimental): Leukemic cells from a patient at relapse can be screened for sensitivity to single compounds
  Interventions: Diagnostic Test: Image-based ex-vivo drug screening platform (pharmacoscopy)

INTERVENTIONS:
Diagnostic Test: Image-based ex-vivo drug screening platform (pharmacoscopy) — Leukemic cells from a patient at relapse can be screened for sensitivity to single compounds. A drug score is calculated for each compound (defined as 1 - (% target cells in drug treated conditions / % target cells under control condition)). If a drug kills all target cells specifically, the best possible score is "1". If the drug is killing all non-target cells, the score goes to negative infinite. If a drug kills both target and non-target cell populations equally, or does nothing, the score is "0".
  Other Names: Pharmacoscopy

SUMMARY:
This is a non-randomised clinical study investigating subsequent patients with specific AML treatment started between January 1, 2022 until December 31, 2022.

Patients with relapsing disease are planned to be analyzed in this study

DETAILED DESCRIPTION:
The standard treatment for young fit patients with acute myeloid leukemia (AML) is intensive chemotherapy followed by consolidation treatment with curative intent. Usually, two cycles of intensive chemotherapy are given, with subsequent consolidation treatment depending on the genetic risk-assessment of the patients as well as on the response to the induction treatment.

For elderly or unfit patients, such an intensive approach is not feasible, and palliative treatment must be considered. The standard first-line-treatment for such patients since more than a decade comprises repetitive cycles of a hypomethylating agent (either Azacitidine or Decitabine). The median progression free survival following these approaches in this population is between 4 and 8 months, with an overall-survival of up to 12 months. More recently, the addition of the Bcl-2 inhibitor Venetoclax to hypomethylating agents has led to a modest improvement both of progression-free and overall survival. However, overall survival in such patients usually does not exceed 14-16 months.

The laboratory of Prof. Berend Snijder, Institute of Molecular Systems Biology, at the ETH (Eidgenössische Technische Hochschule) Zurich has developed an image-based ex-vivo drug screening platform for patients with aggressive haematological malignancies, also called pharmacoscopy. Using such a technique, leukemic cells from a patient at relapse can be rapidly screened for sensitivity to single compounds. A drug score is calculated for each compound.

Starting in Q2/2021, the investigator at the Department of Medical Oncology, University Hospital Inselspital in Bern, collected experiences using such an approach. Having received information from the laboratory on top sensitivity of leukemic cells of a given patient to a specific drug, a process is initiated to try to obtain access to such off-label drugs.

ELIGIBILITY:
Inclusion Criteria:

* Included are patients with AML at relapse treated at the Department of Medical Oncology at the University Hospital Inselspital in Bern.
* Patients are not planned to undergo intensive reinduction treatment with subsequent allogeneic hematopoietic transplantation in a curative intent.
* Patients have exhausted all standard therapeutic options and they must have no available licensed standard treatment for relapsed AML.
* Written informed consent

Exclusion Criteria:

* Patients able to undergo intensive reinduction treatment with subsequent allogeneic hematopoietic transplantation in a curative intent
* Patients have available standard therapeutic options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment with identified effective drug | 12 months
  Percentage of patients with relapsing AML in which drug screening identifies a promising effective drug and in which such a treatment effectively is started

SECONDARY OUTCOMES:
Identification of effective drug | 12 months
  Percentage of patients in which a promising drug can be identified using drug screening
Duration of response | 12 months
  Duration of response of patients effectively treated with a drug identified by drug screening
Overall survival | 12 months
  Overall survival of patients effectively being treated with a drug identified by drug screening.
Response rate of patients depending on the RBF (relative blast fraction) value | 12 months
  Number of patients responding to their chosen therapy regimen in correlation to the RBF (relative blast fraction) value
Duration of response of patients depending on the RBF (relative blast fraction) value | 12 months
  Duration of response in patients responding to their chosen therapy regimen in correlation to the RBF (relative blast fraction) value
Overall survival of patients depending on the RBF (relative blast fraction) value | 12 months
  Overall survival of patients responding to their chosen therapy regimen in correlation to the RBF (relative blast fraction) value

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof Dr. med, Study Chair — Department for Medical Oncology; University Hospital/Inselspital
Locations (1):
- Departement of Medical Oncology, University Hospital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes